CLINICAL TRIAL: NCT02617121
Title: Comparison of the Prophylactic Anti-emetic Efficacy of Gabapentin and Ramosetron in Patients Undergoing Laparoscopic Gynecological Surgery
Brief Title: The Effects of Gabapentin and Ramosetron on Postoperative Nausea and Vomiting in Laparoscopic Gynecological Surgery
Acronym: PONV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HallymUMC
Record Dates: First submitted 2015-11-18; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Gabapentin; ramosetron

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gabapentin (Active Comparator): oral gabapentin 300 mg 1 hours before induction of anesthesia
  Interventions: Drug: Gabapentin
- ramosetron (Active Comparator): ramosetron 0.3 mg iv at end of surgery
  Interventions: Drug: Ramosetron
- Gabapentin and ramosetron (Active Comparator): oral gabapentin 300 mg 1 hours before induction of anesthesia ramosetron 0.3 mg iv at end of surgery
  Interventions: Drug: Gabapentin and Ramosetron

INTERVENTIONS:
Drug: Gabapentin — oral gabapentin 300 mg 1 hour before induction of anesthesia
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Ramosetron — ramosetron 0.3 mg iv at end of surgery
  Other Names: Nasea
  Arms: ramosetron
Drug: Gabapentin and Ramosetron — oral gabapentin 300 mg 1 hour before induction of anesthesia and ramosetron 0.3 mg iv at end of surgery
  Other Names: Neurontin and Nasea
  Arms: Gabapentin and ramosetron

SUMMARY:
This study was designed to compare the effects of gabapentin and ramosetron on PONV in patients undergoing laparoscopic gynecologic surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) in the postanesthesia care unit is a common occurrence after general anesthesia. And laparoscopic gynecological surgery is associated with a high incidence of PONV. Several antiemetic agents such as dopaminergic, histaminic and 5-HT3 antagonist (including ondansetron, ramosetron, granisetron) have been used to prevent PONV. Gabapentin, anti-convulsant, has been shown to decrease PONV, as well as chemotherapy induced nausea and vomiting in recent studies, although the exact mechanism against PONV is not known. The purpose of this study was to compare the efficacy of gabapentin and ramosetron in preventing PONV in patients undergoing laparoscopic gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA physical status 1 and 2 between 20 and 65 years undergoing laparoscopic gynecological surgery with patient-controlled analgesia for postoperative pain control.

Exclusion Criteria:

* Pregnant women
* Patients who took sedatives, antiemetics, hypnotics, analgesics, steroid, or gabapentin
* Patients with neurological deficits
* Patients with history of drug abuse and allergy of study drugs

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | 48 hours postoperative
  The incidence of postoperative nausea and vomiting will be assessed during 48 hours after surgery

SECONDARY OUTCOMES:
Severity of nausea | 48 hours postoperative
  The severity of nausea will be assessed using verbal rating scales (VRS 11-points scales: 0=no nausea to 10=nausea as bad as it could be)
pain score | 48 hours postoperative
  The pain score will be assessed using verbal rating scales (VRS 11-points scales: 0=none to 10=most severe)
sedation score | 48 hours postoperative
  The sedation score will be assessed using verbal rating scales (VRS 11-points scales:0=none to 10=most severe)
patient's overall satisfaction score | 48 hours postoperative
  The patient's overall satisfaction score will be assessed using 5 point scales (5=very satisfied, 4=somewhat satisfied, 3=neither satisfied nor dissatisfied, 2=somewhat dissatisfied, 1=very dissatisfied)
side effects | 48 hours postoperative
  The side effects such as somnolence, dizziness, headache, tremor, diplopia and nystagmus will be assessed and treated

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim KM, Huh J, Lee SK, Park EY, Lee JM, Kim HJ. Combination of gabapentin and ramosetron for the prevention of postoperative nausea and vomiting after gynecologic laparoscopic surgery: a prospective randomized comparative study. BMC Anesthesiol. 2017 May 19;17(1):65. doi: 10.1186/s12871-017-0357-8. PMID 28525981